CLINICAL TRIAL: NCT00231127
Title: Osteoporosis and COPD (Making of a Database)
Brief Title: Osteoporosis and Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Lidwien Graat-Verboom/MD (principal investigator), Catharina Hospital Eindhoven
Other Study IDs: M05-1522
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: COPD; Osteoporosis; Osteopenia
Keywords: COPD; Osteoporosis; Osteopenia; Glucocorticoids; GOLD; BODE
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The goals of the trial are:

* To determine the prevalence of osteoporosis in subgroups of COPD patients.
* To look for risk factors of osteoporosis in COPD patients.
* To create sub-groups for prospective research concerning the effects of bisphosphonates on osteoporosis variables in COPD patients.

DETAILED DESCRIPTION:
Background:

Osteoporosis is defined as a systemically skeletal disorder characterized by a low bone mass and deterioration of the micro-architecture of the bone and is therefore associated with a higher risk of fractures. Large epidemiological studies to determine the incidence and prevalence of osteoporosis in COPD patients in different stages of their disease are not available. The etiology of osteoporosis in COPD patients is complex and depends on multiple factors.

Goals of the Trial:

* To determine the prevalence of osteoporosis in subgroups of COPD patients.
* To look for risk factors of osteoporosis in COPD patients.
* To create sub-groups for prospective research concerning the effects of bisphosphonates on osteoporosis variables in COPD patients.

Study Design:

Patients diagnosed with COPD (according to the American Thoracic Society [ATS] guidelines and divided in stages according to the Global Initiative on Obstructive Lung Diseases [GOLD]-classification) who visit the out-patient clinic of pulmonology of the Catharina Hospital Eindhoven will be asked to participate in the trial. A database will be created (prospectively) of the (medical) information about these patients, which will be analysed retrospective. To gather information we will use the medical records, a questionnaire, a blood sample, long function testing including a 6-minute walking test and a DEXA-scan.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Men and women
* COPD according to the ATS-guidelines, divided in severity according to the GOLD criteria
* Written consent

Exclusion Criteria:

* Age < 18 years
* No written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease Patients visiting the pulmonary outpatient clinic of the Catharina Hospital Eindhoven.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2005-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lidwien Graat, MD, Principal Investigator — Catharina Hospital Eindhoven (Department of Pulmonology)
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, North Brabant, Netherlands